CLINICAL TRIAL: NCT01899547
Title: Laparoscopy-Assisted Surgery for Carcinoma of the Low Rectum : A Prospective, Multi-Center, Randomized, Open-Label, Parallel Group, Non-Inferiority Clinical Trial
Brief Title: Laparoscopy-Assisted Surgery for Carcinoma of the Low Rectum
Acronym: LASRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other); Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other); Liaoning Cancer Hospital & Institute (Other); RenJi Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other); Shengjing Hospital (Other); Fujian Cancer Hospital (Other Government); The Second Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Longyan Affiliated Hospital, Fujian Medical University (Unknown); Fudan University (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-sen University (Other); Hubei Cancer Hospital (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Pan Chi, MD, Chief of Department of General Surgery, Fujian Medical University Union Hospital, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0925-0586; LASRE (Registry Identifier: Laparoscopy-assisted Surgery for Carcinoma of the Low Rectum)
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo laparoscopic-assisted rectal resection.
  Interventions: Procedure: laparoscopic-assisted rectal resection
- Arm II (Active Comparator): Patients undergo conventional open rectal resection.
  Interventions: Procedure: conventional open rectal resection

INTERVENTIONS:
Procedure: laparoscopic-assisted rectal resection — Arm I: Patients undergo laparoscopic-assisted rectal resection.
  Arms: Arm I
Procedure: conventional open rectal resection — Arm II: Patients undergo conventional open rectal resection.
  Arms: Arm II

SUMMARY:
The purpose of this study is to evaluate the safety and oncological feasibility of laparoscopy-assisted surgery for low rectal carcinoma compared with open surgery.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven rectal adenocarcinoma
* inferior edge of the tumor located within 5 cm from the dentate line as determined by rigid proctoscopy
* diagnosis of rectal cancer amenable to curative surgery either by anterior resection or abdominoperineal resection or extralevator abdominoperineal excision
* T3-4a,N0 or T1-4a,N1-2 treated with neoadjuvant chemoradiotherapy
* no evidence of distant metastases
* tumor size <6cm
* sufficient organ function
* no contraindication to laparoscopic surgery
* without other malignancies in medical history

Exclusion Criteria:

* concurrent or previous diagnosis of invasive cancer within 5 years
* locally advanced cancers requiring en bloc multivisceral resection
* intestinal obstruction
* intestinal perforation
* history of colorectal surgery
* American Society of Anesthesiologists(ASA) class 4 or 5
* pregnant or breast-feeding women
* history of mental disorder
* participation in another rectal cancer clinical trial relating to surgical technique

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
3 years disease-free survival | 3 years
  Disease-free survival is defined as the time from date of surgery to the date of rectal cancer recurrence or metastasis or cancer-related death (locoregional or distant recurrence) .

SECONDARY OUTCOMES:
Pathologic outcomes | 1 week post operatively
  Pathologic outcomes are defined as TME quality, negative CRM and negative DRM, length of proximal resection margin (PRM), length of DRM, and the number of retrieved lymph nodes.The TME quality was graded based on the criteria proposed by Nagtegaal et al. as complete, nearly complete, or incomplete.Positive resection margin, including circumferential resection margin (CRM) and distal resection margin (DRM), was defined as the presence of cancer cells within 1 mm from the cut edge.
30-day postoperative complications | 1 month within operatively
  Thirty-day postoperative complications included any complications occurring within 30 days after surgery. Postoperative complications were graded according to the Clavien-Dindo classification. Severe complications were defined as Clavien-Dindo III-V.
30-day postoperative mortality | 30 days post operatively
  Thirty-day operative mortality is defined as deaths occurring from any cause during the first 30 postoperative days.
Overall survival | 3 and 5 years post operatively
  Overall survival is defined as the time from date of surgery to date of death from any cause.
Locoregional recurrence rate | 3 and 5 years post operatively
  Locoregional recurrence was defined as the presence of any anastomotic, pelvic or perineal tumour documented by clinical and/or pathological examination.

OTHER OUTCOMES:
Operative time | Day 1
  Operative time is defined as the time from skin incision to the completion of skin suture.
Conversion to Open Surgery | Day 1
  The conversion is defined as any part of the mesorectal dissection using the traditional open surgery. The surgeon decided the conversion after considering patient safety, technical difficulties, and relevant conditions influencing the completion of TME.
Estimated blood loss | Day 1
  Estimated blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
Length of hospital stay | from the completion of the surgery till discharge from hospital
  Duration of hospital stay measured from the day of surgery until the day of discharge from hospital.
Patient self-reported bladder and sexual function | at postoperative 3,6 and 12 months
  Patient self-reported bladder and sexual function as assessed by the International Prostatic Symptom Score(I-PSS©) for male and female bladder function and the International Index of Erectile Function (IIEF) Female Sexual Function Index(FSFI©) for sexual function.
Health related quality of life | at postoperative 3,6 and 12 months
  Health related quality of life assessed by EORTC CR29 score, EORTC CR30 score

CONTACTS AND LOCATIONS:
Overall Officials: Pan Chi, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Sun Y, Tang Z, Jiang W, Wang X, Huang Y, Chi P. Textbook outcome in low rectal cancer patients undergoing laparoscopic or open surgery: 3-year results from the multicentric LASRE Trial. Int J Colorectal Dis. 2025 Aug 13;40(1):177. doi: 10.1007/s00384-025-04976-w. PMID 40804342
- [Derived] Jiang W, Xu J, Cui M, Qiu H, Wang Z, Kang L, Deng H, Chen W, Zhang Q, Du X, Yang C, Guo Y, Zhong M, Ye K, You J, Xu D, Li X, Xiong Z, Tao K, Ding K, Zang W, Feng Y, Pan Z, Wu A, Huang F, Huang Y, Wei Y, Su X, Chi P; LASRE trial investigators. Laparoscopy-assisted versus open surgery for low rectal cancer (LASRE): 3-year survival outcomes of a multicentre, randomised, controlled, non-inferiority trial. Lancet Gastroenterol Hepatol. 2025 Jan;10(1):34-43. doi: 10.1016/S2468-1253(24)00273-5. Epub 2024 Nov 8. PMID 39527970
- [Derived] Jiang WZ, Xu JM, Xing JD, Qiu HZ, Wang ZQ, Kang L, Deng HJ, Chen WP, Zhang QT, Du XH, Yang CK, Guo YC, Zhong M, Ye K, You J, Xu DB, Li XX, Xiong ZG, Tao KX, Ding KF, Zang WD, Feng Y, Pan ZZ, Wu AW, Huang F, Huang Y, Wei Y, Su XQ, Chi P; LASRE trial investigators. Short-term Outcomes of Laparoscopy-Assisted vs Open Surgery for Patients With Low Rectal Cancer: The LASRE Randomized Clinical Trial. JAMA Oncol. 2022 Sep 15;8(11):1607-15. doi: 10.1001/jamaoncol.2022.4079. Online ahead of print. PMID 36107416
- [Derived] Chi P. [Laparoscopic total mesorectum excision with the guidance of membrane anatomy]. Zhonghua Wei Chang Wai Ke Za Zhi. 2016 Oct 25;19(10):1088-1091. Chinese. PMID 27781241